CLINICAL TRIAL: NCT03732898
Title: Coordinated Reset Deep Brain Stimulation (RESET-DBS) and RESET-DBS - Extension (Sub-study)
Brief Title: Coordinated Reset Deep Brain Stimulation
Acronym: RESET-DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A4058
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: During follow-up, the conventional Deep Brain Stimulation (cDBS) program and one or more of these novel Deep Brain Stimulation (nDBS) programs are programmed into a subject's IPG. At the investigator's discretion, a copy of the cDBS program may also be stored in one of the investigational slots. The subject will be blinded to the slot number assignment for the cDBS program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Novel Deep Brain Stimulation (nDBS) program (Experimental): This arm will include patients receiving stimulation with a novel Deep Brain Stimulation (nDBS) for Parkinson's Disease (PD).
  Interventions: Device: Novel Programming (nDBS)
- Conventional Deep Brain Stimulation (cDBS) program (Active Comparator): This arm will include patients receiving stimulation with a conventional Deep Brain Stimulation (cDBS) for Parkinson's Disease (PD).
  Interventions: Device: Conventional Programming (cDBS)

INTERVENTIONS:
Device: Novel Programming (nDBS) — The commercial CP installed with the investigational DBS programming software will be used to set up Novel Programming (nDBS) therapy on the IPG.
  Arms: Novel Deep Brain Stimulation (nDBS) program
Device: Conventional Programming (cDBS) — The commercial CP installed with commercial software will be used to set up standard cDBS therapy on the IPG.
  Arms: Conventional Deep Brain Stimulation (cDBS) program

SUMMARY:
The study will explore the viability of an alternative/novel programming strategy in Deep Brain Stimulation (DBS) for patients with Parkinson's Disease (PD).

DETAILED DESCRIPTION:
The study will explore the feasibility of utilizing an alternative/novel programming technique in Deep Brain Stimulation (DBS) for patients with Parkinson's Disease (PD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject with PD implanted bilaterally in the STN and receiving DBS therapy for at least 3 months.
2. Tolerates > 12 hours OFF medication and, per clinical judgment, be able to perform all study related procedures.
3. Able to understand the study requirements and the treatment procedures and must provide written informed consent before any study-specific tests or procedures are performed.

Key Exclusion Criteria:

1. Exhibits significant psychiatric problems, including unrelated clinically significant depression as determined by the investigator.
2. A female who is pregnant, is breastfeeding, or is of childbearing potential and planning to get pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Quality of Life using new programming paradigm: PDQ-39 | approximately 4 weeks
  Change in Parkinson's Disease Questionnaire (PDQ-39) summary index and sub-scores

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Neuromodulation Corporation
Locations (2):
- Germany (2):
  - University Berlin, Charite Virchow, Berlin
  - Universitaetsklinikum Wuerzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No